CLINICAL TRIAL: NCT00696618
Title: A Randomized, Blinded, Comparative Study of the Mucosal Toxicity, Colorectal Distribution, and Participant Acceptability of Three Different Preparatory Enemas (Hypo-, Iso-, and Hyper-osmolar)
Brief Title: Enema Use and Acceptability in HIV Negative Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00010972
Record Dates: First submitted 2008-06-04; First posted 2008-06-13 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
Keywords: HIV prevention; MSM; Enema; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — sodium phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Tap water enema (hypo-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 1), Followed by Normosol-R enema (iso-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home(Stage 2), Followed by Fleet enema (hyper-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 3)
  Interventions: Drug: Fleet Enema; Drug: tap water enema; Drug: Normosol-R enema
- B (Experimental): Normosol-R enema (iso-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 1), Followed by Fleet enema (hyper-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 2), Followed by Tap water enema (hypo-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 3)
  Interventions: Drug: Fleet Enema; Drug: tap water enema; Drug: Normosol-R enema
- C (Experimental): Fleet enema (hyper-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 1), Followed by Tap water enema (hypo-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 2), Followed by Normosol-R enema(iso-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 3)
  Interventions: Drug: Fleet Enema; Drug: tap water enema; Drug: Normosol-R enema

INTERVENTIONS:
Drug: Fleet Enema — hyper-osmolar preparation
  Other Names: hyperosmolar enema
Drug: tap water enema — hypo-osmolar preparation
  Other Names: hypo-osmolar enema
Drug: Normosol-R enema — iso-osmolar preparation
  Other Names: iso-osmolar enema

SUMMARY:
This study is looking at 3 different types of enemas used before receptive anal intercourse in men who have sex with men (MSM). We are investigating whether the enemas cause any damage to the lining of the colon, how far up the colon the enemas travel after they are given, and how much study participants like using each of the enemas.

DETAILED DESCRIPTION:
Research participants who are deemed eligible after screening will return for a baseline evaluation. The baseline visit includes clinical evaluation and colon tissue collection, as well as a Baseline Behavioral Questionnaire (BBQ). The BBQ will be administered by Computer Assisted Self-Interview (CASI). Participants may complete the web-based CASI in the privacy of their own home.

Following the baseline visit, participants will be randomized into one of three groups. Each group will receive enemas of varying osmolality (molecule concentrations) in a different sequence according to study stage. During each stage of enema test product use participants will receive a single inpatient dose followed by three outpatient doses to be used in the context of Receptive Anal Intercourse (RAI).

This study will involve 3 stages of enema test product use. Each stage is identical, with the exception of the enema osmolality. Each stage includes an inpatient period and an outpatient period. The time period between stages 1, 2, and 3 will be approximately 2-6 weeks to allow for a recovery period, opportunities for product use, and appointment availability. The participant's inpatient portion of the study will take place as scheduling permits after the at-home enema use is complete.

During each stage, the participant is admitted to the inpatient unit for <48 hours, placed on a clear liquid diet, and has an interval medical history and directed physical exam. The following day the 125ml study enema is radiolabeled and administered to the participant. Over an approximately 25 hour time period, the participant will undergo pharmacokinetic studies involving blood drawing, colon tissue sample collection by flexible sigmoidoscopy, and imaging by Single Photon Emission Computed Tomography/ paired with x-ray Computed Tomography (SPECT/CT). The participant will then be discharged home with 3 doses of study enema. Participants will be instructed to allow for an approximately 72 hour recovery period (to ensure healing of the colon tissue biopsy sites) prior to initiating use of the study product on an outpatient basis, if applicable. Subjects will be encouraged to use the study product on 3 separate occasions in the context of RAI. As with standard HIV counseling, participants will be encouraged to use condoms. After each outpatient use the subject will complete a Brief Acceptability Questionnaire (BAQ). Then at the end of each stage of enema test article use, the subject will complete a Product Acceptability Questionnaire (PAQ).

Study Exit Interview At completion of all 3 stages the participant will complete an Overall Product Preference Questionnaire (OPPQ) administered by CASI followed by and in-depth interview.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥ Age of 18
* HIV-1 status antibody negative as documented at screening
* A history of RAI at least twice per month in the prior 3 months*

  * Required to assure that subjects are likely to complete each stage of enema test article use in a reasonable amount of time.
* History of enema use prior to RAI at least some of the time
* Willing to use each study product prior to RAI on 3 separate occasions.
* Willing to refrain from RAI for 48 hours before and after inpatient periods.
* Willing to use condoms for the duration of the study
* Availability to return for all study visits, barring unforeseen circumstances
* Understands and agrees to local Sexually Transmitted Infection (STI) reporting requirements
* Able and willing to communicate in English
* Able and willing to provide written informed consent to take part in the study
* Able and willing to provide adequate information for locator purposes

Exclusion Criteria:

* Female
* HIV positive at baseline
* History of inflammatory bowel disease
* Active inflammatory condition of the GI tract at baseline
* Active rectal infection at Visit 2 (Infections identified during the screening period must be treated prior to Visit 2)
* Presence of any painful anorectal conditions that would be tender to manipulation. (Participants with hemorrhoids and/or anal warts that are not painful may participate.)
* History of prosthetic cardiac valves, including bioprosthetic and homograft valves, previous bacterial endocarditis, surgically constructed systemic pulmonary shunts or conduits, and complex cyanotic congenital heart disease such as single ventricle states, transposition of the great arteries, tetralogy of Fallot or similar conditions that put the subject at high risk for bacteremia during endoscopy, hence requiring antibiotic prophylaxis.
* Unwillingness to refrain from chronic use of aspirin and NSAIDs.
* Use of warfarin or heparin
* Use of systemic immunomodulatory medications within 72 hours of Visit 2 baseline
* Use of rectally administered medications, including over-the-counter enemas, within 72 hours of Visit 2 baseline
* Use of product containing nonoxynol-9 rectally within 72 hours of Visit 2
* Use of any investigational products within 72 hours of Visit 2 baseline
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral disease, or coagulopathies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited to the outpatient clinical unit via a volunteer screening database.Similarly, individuals may have responded to advertisements posted throughout the Johns Hopkins Medical Institutions or via word of mouth from other research participants. Individuals were recruited between 10/10/07 and 01/06/09.
Pre-assignment Details: Seventeen subjects were recruited. Eight individuals did not meet screening criteria and were not enrolled.
Groups:
- Tap Water/Normosol-R/Fleet: Tap water enema (hypo-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 1), Followed by Normosol-R enema (iso-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home(Stage 2), Followed by Fleet enema (hyper-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 3)
  Fleet Enema: hyper-osmolar preparation
  tap water enema: hypo-osmolar preparation
  Normosol-R enema: iso-osmolar preparation
- Normosol-R/Fleet/Tap Water: Normosol-R enema (iso-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 1), Followed by Fleet enema (hyper-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 2), Followed by Tap water enema (hypo-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 3)
  Fleet Enema: hyper-osmolar preparation
  tap water enema: hypo-osmolar preparation
  Normosol-R enema: iso-osmolar preparation
- Fleet/Tap Water/Normosol-R: Fleet enema (hyper-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 1), Followed by Tap water enema (hypo-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 2), Followed by Normosol-R enema(iso-osmolar) administered rectally 125 mL one time in the clinic, then self-administered on three separate occasions at home (Stage 3)
  Fleet Enema: hyper-osmolar preparation
  tap water enema: hypo-osmolar preparation
  Normosol-R enema: iso-osmolar preparation
Period: Overall Study
Arm/Group | Tap Water/Normosol-R/Fleet | Normosol-R/Fleet/Tap Water | Fleet/Tap Water/Normosol-R
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tap Water/Normosol-R/Fleet | Normosol-R/Fleet/Tap Water | Fleet/Tap Water/Normosol-R | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mucosal Toxicity Using Histopathology
Description: Endoscopy will be performed to obtain biopsy specimens at baseline and following each inpatient enema exposure. Samples will be obtained at each flexible sigmoidoscopy and set aside for batch sectioning and H&E staining. Slides will be reviewed and scored by a qualified pathologist blinded to treatment assignment using a qualitative scoring system. This scoring system uses semi-quantitative scoring that focuses on acute toxicity to epithelial cell layer similar to that seen in animal studies. This is a categorical grading scale, where 0 = Epithelial surface intact;1 = <1/3 of surface denuded; 2 = 1/3 - 2/3rds of surface denuded;3 = More than 2/3rds of surface denuded.
  Six separate biopsies for each subject and each treatment intervention were analyzed in a multi-level analysis. In comparison with the baseline condition (no intervention), the odds and 95% confidence interval (CI) of having a higher epithelial denudation score were calculated for each intervention.
Time Frame: One hour following enema exposure
Population: All participants who received one dose of each intervention and completed all study visits were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: colon biopsies
Groups:
- Hypo-osmolar Enema: Hypo-osmolar Tap water enema
- Iso-osmolar Enema: Normosol-R Iso-osmolar enema
- Hyper-osmolar Enema: Fleet Hyper-osmolar enema
Arm/Group | Hypo-osmolar Enema | Iso-osmolar Enema | Hyper-osmolar Enema
Number analyzed (Participants) | 9 | 9 | 9
Number analyzed (colon biopsies) | 54 | 54 | 54
units on a scale | 0.6 [0.2 to 1.7] | 0.5 [0.2 to 1.5] | 4.2 [1.7 to 10.1]
Statistical Analysis 1: Comparison: Hypo-osmolar Enema vs Iso-osmolar Enema vs Hyper-osmolar Enema; Nine research participants provided the ability to detect an effect size of 1.25 standard deviation units relative to the mean with 80% power using two-sided, 5% alpha in a paired analysis. The Baseline condition (no intervention) was assigned a value of 1 and geometric mean ratios with 95% confidence intervals for each intervention were calculated relative to baseline; Test type: Superiority or Other; p < .05, multi-level — Adjusted for multiple comparisons

2. Secondary Outcome: Radiolabel Area Under the Curve (AUC 0-24 hr)
Description: Percent of radiolabel dose administered was determined by plasma sampling at standardized intervals over 24 hours. AUC was then calculated using the trapezoidal rule and reported as x10 log 7 microcurie-hours/mL
Time Frame: 24 hours following each intervention
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 10 log 7 microcurie-hours/mL
Arm/Group | Hypo-osmolar Enema | Iso-osmolar Enema | Hyper-osmolar Enema
Number analyzed (Participants) | 9 | 9 | 9
10 log 7 microcurie-hours/mL | 21.4 [17.4 to 44.9] | 19.7 [8.4 to 27.4] | 9.4 [8.7 to 13]
Statistical Analysis 1: Comparison: Hypo-osmolar Enema vs Iso-osmolar Enema vs Hyper-osmolar Enema; Test type: Superiority or Other; p < .05, multi-level

3. Secondary Outcome: D(Average) at Two Hours
Description: Mean proximal residence distance of radio-signal from anus as measured on SPECT/CT
Time Frame: two hours following dosing of intervention
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: centimeters
Arm/Group | Hypo-osmolar Enema | Iso-osmolar Enema | Hyper-osmolar Enema
Number analyzed (Participants) | 9 | 9 | 9
centimeters | 8.6 [6.8 to 11.8] | 20.6 [17.4 to 25.6] | 7.7 [0 to 14.4]
Statistical Analysis 1: Comparison: Hypo-osmolar Enema vs Iso-osmolar Enema vs Hyper-osmolar Enema; Test type: Superiority or Other; p < .05, mulit-level analysis

ADVERSE EVENTS:
Arm/Group | Hypo-osmolar Enema | Iso-osmolar Enema | Hyper-osmolar Enema
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 2/9 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypo-osmolar Enema (N=9) | Iso-osmolar Enema (N=9) | Hyper-osmolar Enema (N=9)
Procedure-related (Investigations) | 4 (7) | 2 (3) | 3 (5) — adverse events secondary to study procedures, including musculoskeletal complaints from positioning in scanner, bloating/gas following endoscopy, hematoma from blood drawing.
GI complaints thought related to study product (Product Issues) | 0 (0) | 1 (1) | 1 (1) — Includes lower GI complaints such as rectal tenderness, anal canal irritation
GI complaints other (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) — Includes other GI disorders not believed to be related to study product (E.g. nausea/vomiting, diarrhea related to intercurrent illness)
Dizzyness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial cut (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No